CLINICAL TRIAL: NCT00001349
Title: Apheresis Procedures to Obtain Plasma or Leukocytes for In Vitro Studies
Brief Title: Apheresis to Obtain Plasma or White Blood Cells for Laboratory Studies
Status: Terminated | Type: Observational
Why Stopped: Closed at the request of the IRBO
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930057; 93-I-0057
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Leukopheresis; Plasmapheresis
Keywords: Plasmapheresis; Lymphocytes; Eosinophils; Neutrophils

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Leukocytes, platelets and plasma will be collected. Since this protocol only allows for apheresis to be performed on participants enrolled on another LPD protocol, any biological samples collected will be covered by the other, individual protocol on which the participant is enrolled.

GROUPS / COHORTS (1):
- 1: Donors first admitted to another approved clinical research protocol of the NIAID before having the apheresis procedures described in this protocol.

SUMMARY:
This study will collect blood plasma and white blood cells for laboratory research using a procedure called apheresis. Apheresis is a method of collecting larger quantities of certain blood components than can safely be collected through a simple blood draw.

Patients 7 years of age and older with a parasitic infection or condition associated with a parasitic infection (i.e., elevated levels of IgE antibodies or of a type of white cell called eosinophils) who are currently enrolled in a NIH clinical research protocol may be eligible for this study. Relatives of patients and normal healthy volunteers will also be enrolled. Candidates will have a medical history, physical examination and blood tests. Individuals weighing less than 25 kilograms (55 pounds) may not participate.

Participants will undergo one of the following two apheresis procedures:

* Automated pheresis Whole blood is drawn through a needle placed in an arm vein and circulated through a cell separator machine. The plasma (liquid part of the blood) and white cells are extracted, and the red cells are re-infused into the donor through a needle in the other arm. The procedure takes 1 to 2 hours.
* Manual pheresis Whole blood is drawn through a needle placed in an arm vein and circulated through the cell separator machine. The red blood cells are separated from the rest of the blood and returned to the donor through the same needle. Usually only one needle stick is required and the procedure takes from 30 to 45 minutes. This method is used only in individuals who weigh less than 35 kg (77 pounds).

DETAILED DESCRIPTION:
In order to carry out in vitro research procedures on the plasma or leukocyte components of blood, it is often necessary to obtain larger quantities of plasma and/or leukocytes, than can be safely obtained by simple phlebotomy. These components can be easily and safely obtained using apheresis procedures in the Clinical Center Apheresis Unit. This protocol is specifically designed to conform to the requirements of the Apheresis Unit for donors to have apheresis procedures (>7 years of age and greater than or equal to 25kg). Donors must first be admitted to another approved clinical research protocol of the LPD, NIAID before they may have the apheresis procedures described in this protocol. The investigational nature of the studies in which the samples will be used, as well as the risks and benefits of the donation process will be explained to all donors, and a signed informed consent document will be obtained.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Enrolled on another LPD protocol.
* Weight greater than or equal to 25 kg
* Willingness to participate

EXCLUSION CRITERIA:

* Age less than 7 years
* Weight less than 25 kg
* Cardiovascular instability
* Hct less than 30
* Inadequate venous access
* PTT or PT greater than 1.5 normal
* Pregnancy
* Women who are actively breastfeeding
* Other condition which the attending physician or Apheresis Unit staff considers a contraindication to the procedure
* For Hetastarch procedure

  * Hypertension
  * Evidence of fluid retention

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any subject enrolled on an existing !RB-approved LPD protocol may be asked to participate and thereby undergo apheresis.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Actual)
Dates: Start 1993-03-23 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
To obtain leukocytes,platelets, and plasma from subjects already enrolled on other NIAID/LPD protocols. | Ongoing as this is a method to collect cells from subjects enrolled on other LPD protocols
  Leukocytes, platelets, and plasma will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas B Nutman, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Boyd A, Ribeiro JM, Nutman TB. Human CD117 (cKit)+ innate lymphoid cells have a discrete transcriptional profile at homeostasis and are expanded during filarial infection. PLoS One. 2014 Sep 25;9(9):e108649. doi: 10.1371/journal.pone.0108649. eCollection 2014. PMID 25255226
- [Background] Chatterjee S, Clark CE, Lugli E, Roederer M, Nutman TB. Filarial infection modulates the immune response to Mycobacterium tuberculosis through expansion of CD4+ IL-4 memory T cells. J Immunol. 2015 Mar 15;194(6):2706-14. doi: 10.4049/jimmunol.1402718. Epub 2015 Feb 9. PMID 25667413
- [Background] Santiago Hda C, Ribeiro-Gomes FL, Bennuru S, Nutman TB. Helminth infection alters IgE responses to allergens structurally related to parasite proteins. J Immunol. 2015 Jan 1;194(1):93-100. doi: 10.4049/jimmunol.1401638. Epub 2014 Nov 17. PMID 25404363
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1993-I-0057.html